CLINICAL TRIAL: NCT00113204
Title: A Phase 1, Safety Assessment and Pharmacokinetic Study of IPI-504 in Patients With Relapsed, and Relapsed Refractory Multiple Myeloma
Brief Title: Safety Study of IPI-504 in Patients With Relapsed and Relapsed Refractory Multiple Myeloma
Acronym: IPi-504-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-01
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Relapsed; Relapsed refractory; Hematologic cancer; hematologic disease; plasma cells
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Hematologic Neoplasms; Hematologic Diseases | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IPI-504

SUMMARY:
This is a phase 1 clinical trial to find the safe, maximum tolerated dose of IPI-504 in patients with relapsed and/or relapsed, refractory multiple myeloma. This study will examine how IPI-504 is absorbed, distributed, metabolized, and eliminated by the body. The study will also evaluate potential anti-tumor activity of IPI-504.

DETAILED DESCRIPTION:
IPI-504 is a novel small molecule inhibitor of heat shock protein 90 (Hsp90), an emerging and recently identified target for cancer therapy. Hsp90 is a protein chaperone that plays a central role in regulating protein homeostasis. Hsp90 regulates the stability of key proteins (called "client proteins") and keeps them in the appropriate three dimensional shape so they can perform their cellular functions. In addition, many of the proteins stabilized by Hsp90 are oncoproteins and cell-signaling proteins important in cancer cell proliferation and cancer cell survival. Thus Hsp90, a single molecular target that is a central integrator of multiple pathways important to cancer, is an ideal novel target for oncologic therapy. Selective inhibition of Hsp90 will affect multiple downstream mechanisms to disrupt tumor growth and selectively kill cancer cells. The anti-neoplastic effects of Hsp90 inhibition have been demonstrated both in vitro and in vivo for a variety of different hematologic and solid tumors including multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or relapsed, refractory disease
* Age is greater or equal to 18 years at the time of signing the informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Ability to adhere to the study visit schedule and all protocol requirements
* Voluntarily sign an informed consent
* All baseline studies must be completed for determining eligibility within 21 days of study enrollment
* Women of child-bearing potential (WCBP) defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post-menopausal for at least 24 consecutive months must have a negative serum or urine pregnancy test prior to each cycle of treatment
* All WCBP and all sexually active male patients must agree to use adequate methods of birth control throughout the study

Exclusion Criteria:

* Disease specific treatment within the previous 3 weeks including use of chemotherapy that is known to be active or may be active against multiple myeloma
* Previous treatment with 17-AAG, DMAG, or other known Hsp90 inhibitor
* Participation in any investigational drug study within 3 weeks preceding start of treatment for conventional small molecule therapy or 4 weeks preceding the start of treatment for biologic or vaccine therapy; concurrent radiation therapy is not permitted
* Concomitant use of corticosteroids may not exceed prednisone 10 mg per day with the exception of pre-medication for transfusion of blood products and topical application
* Concurrent treatment with any agent that alters CYP3A activity (unless maintained on stable dose)
* Baseline QTc >450
* NYHA class 3 or 4 congestive heart failure
* Left Bundle Branch Block
* Mycardial infarction or active ischemic heart disease within 6 months
* Grade 3 or greater peripheral neuropathy
* Renal insufficiency, serum creatinine >2x upper limit of normal (ULN)
* Platelets < 30,000 mm3 or refractory to transfusion and unable to be maintained > 50,000 mm3
* AST and / or ALT > 2.0x ULN
* ANC <1,000 cells/mm3
* Hemoglobin < 8.0 g/dL
* Presence of active infection or systemic use of antibiotics within 72 hours of treatment
* WCBP who are breast feeding
* Significant co-morbid condition or disease which in the judgment of the investigator would place the patient at undue risk or interfere with the study (e.g. cardiac disease such as acute coronary syndrome or unstable angina within 6 months, New York Heart Association (NYHA) class 2 or greater congestive heart failure (CHF), uncontrolled hypertension, arrhythmia requiring medication or mechanical control, chronic obstructive pulmonary disease (COPD), cirrhotic liver disease, or other conditions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety and maximum tolerated dose of IPI-504 | Following 1 cycle of treatment
Recommend a dose for subsequent studies of IPI-504 | Once MTD is reached

SECONDARY OUTCOMES:
To examine the pharmacokinetic parameters of IPI-504 | During first dose first cycle of IPI-504
To evaluate the potential anti-tumor activity with standard markers of disease progression | 1 cycle of treatment
To examine pharmacodynamic markers of biologic activity of IPI-504 | Cycle 1 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Jagannath, MD, Principal Investigator — St. Vincent's Comprehensive Cancer Center; David S. Siegel, MD; Ph.D, Principal Investigator — Hackensack Meridian Health; Ivan Borrello, MD, Principal Investigator — Johns Hopkins - Sidney Kimmel Comprehensive Cancer Center; Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center The David Jurist Research Center, Hackensack, New Jersey
  - St. Vincent's Comprehensive Cancer Center, New York, New York

REFERENCES:
- [Background] Maloney A, Workman P. HSP90 as a new therapeutic target for cancer therapy: the story unfolds. Expert Opin Biol Ther. 2002 Jan;2(1):3-24. doi: 10.1517/14712598.2.1.3. PMID 11772336
- [Background] Pratt WB, Toft DO. Regulation of signaling protein function and trafficking by the hsp90/hsp70-based chaperone machinery. Exp Biol Med (Maywood). 2003 Feb;228(2):111-33. doi: 10.1177/153537020322800201. PMID 12563018
- [Background] Neckers L. Hsp90 inhibitors as novel cancer chemotherapeutic agents. Trends Mol Med. 2002;8(4 Suppl):S55-61. doi: 10.1016/s1471-4914(02)02316-x. PMID 11927289
- See also: Click here for more information about Multiple Myeloma — http://www.multiplemyeloma.org/